CLINICAL TRIAL: NCT07233538
Title: Effect of Preoperative Ultrasound-guided Bilateral Maxillary Nerve Block Via the Pterygopalatine Fossa on Intraoperative Remifentanil Use in Septorhinoplasty
Brief Title: Preoperative Maxillary Nerve Block and Remifentanil Use in Septorhinoplasty
Acronym: PRISM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Can Ozan Yazar, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AEŞH-EK-2025-191
Record Dates: First submitted 2025-08-06; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Surgery; Plastic Surgery; Rhinoplasty; Pain; Regional Anaesthesia; Nerve Blocks
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Maxillary (Active Comparator): Maxillary block group And General Anesthesia
  Interventions: Procedure: Maxillary block
- Group control (No Intervention): Only General Anesthesia

INTERVENTIONS:
Procedure: Maxillary block — Bilateral maxillary nerve block in the preoperative phase
  Arms: Group Maxillary

SUMMARY:
Septorhinoplasty is generally a prolonged surgical procedure that frequently involves osteotomy, which may lead to increased intraoperative remifentanil requirements. Moreover, it is often associated with significant bleeding due to the dense capillary network of the nasal region, making the maintenance of low-to-normal blood pressure preferable during surgery. Consequently, achieving stable hemodynamics and providing sufficient analgesia throughout the procedure is essential.

This study aims to evaluate the effects of bilateral maxillary nerve block on intraoperative remifentanil consumption and postoperative analgesic efficacy in patients undergoing Septorhinoplasty. A total of 90 patients will be included in the study. Forty-five patients (Group M) will undergo Septorhinoplasty under general anesthesia combined with bilateral maxillary nerve block, while the remaining 45 patients (Group N) will receive general anesthesia alone.

In the preoperative phase, a bilateral maxillary nerve block will be performed under ultrasound guidance via the pterygopalatine fossa. During the intraoperative period, total remifentanil consumption will be recorded, alongside assessments of hemodynamic stability, sevoflurane consumption, extubation time, intraoperative bleeding volume, and the satisfaction levels of both the anesthesiologist and the surgeon.

In the postoperative period, patient satisfaction, pain scores at 0, 1, 2, 4, 6, 12, 18, and 24 hours as well as at 1 month (measured using the Visual Analog Scale - VAS), additional analgesic requirements, and Quality of Recovery-15 (QoR-15) scores (assessed on preoperative day 1, postoperative day 1, and at 1 month) will be evaluated.

DETAILED DESCRIPTION:
Septorhinoplasty is a surgical procedure that involves reshaping the nasal soft tissues, cartilage, and bone, and it frequently requires osteotomy. Manipulation of these structures typically results in moderate to severe postoperative pain. Nearly 30% of patients report pain scores of 6 or higher on the Numeric Rating Scale (NRS). Additionally, the use of nasal tampons in the postoperative period may exacerbate discomfort.

For postoperative pain management, nonsteroidal anti-inflammatory drugs (NSAIDs) and opioids may be used. The American Society of Anesthesiologists (ASA) recommends the use of multimodal analgesia combined with regional anesthesia techniques during the perioperative period for the management of acute pain. The incorporation of regional techniques enhances analgesic efficacy synergistically and helps reduce opioid requirements, thereby lowering the incidence of related adverse effects. Moreover, regional techniques applied in the preoperative period are known to support more stable hemodynamic responses.

The trigeminal nerve provides the primary sensory innervation of the face. Its maxillary branch (V2) innervates the nasopharynx, palate, nasal cavity, maxillary sinus, skin of the nasal sidewall, and upper lip. After exiting the middle cranial fossa, it passes through the foramen rotundum and enters the pterygopalatine fossa, where it gives rise to several sensory branches. Among these, the infraorbital and nasopalatine nerves supply sensory innervation to the nasal septum mucosa. The posterior, superior, and inferior lateral nasal nerves, which also arise from the maxillary nerve, innervate the superior, middle, and inferior turbinates. Other branches supply sensation to the skin of the nasal ala and upper lip.

Although bilateral isolated infraorbital nerve block-a branch of the maxillary nerve-has been shown to provide analgesia following nasal surgeries, several studies have reported that analgesia may remain insufficient even with the addition of an infratrochlear nerve block. Therefore, rather than targeting individual branches, blockade of the maxillary nerve itself has been proposed. For this purpose, ultrasound-guided injection via the pterygopalatine fossa has been described.

The aim of this study is to compare intraoperative remifentanil consumption between patients who receive a preoperative bilateral maxillary nerve block and those who do not.

The investigators hypothesize that bilateral maxillary nerve block provides effective intraoperative analgesia, reduces remifentanil requirements, and ensures adequate postoperative pain control.

A total of 90 patients will be enrolled. Randomization will be conducted using the closed-envelope method. The anesthesiologist performing the block and the anesthesiologist responsible for intraoperative and postoperative management will be different individuals, with the latter blinded to group allocation. Patients who receive the block will be assigned to Group M, while those who do not will be assigned to Group N. Group allocation will remain concealed from all personnel except the anesthesiologist administering the block and the study investigators.

All patients will undergo surgery under general anesthesia. A preoperative fasting period of 8 hours for both solids and liquids will be required. Upon admission to the preoperative observation clinic, noninvasive blood pressure (NIBP) and heart rate (HR) will be measured. The average preoperative NIBP and HR values will be calculated based on the last two recordings obtained in the ward. The Quality of Recovery-15 (QoR-15) questionnaire will also be administered at this time.

In the designated block area of the preoperative care unit, patients in Group M will receive a bilateral maxillary nerve block with 4 mL of 0.5% bupivacaine on each side (total volume: 8 mL). Following administration, patients will be monitored for 30 minutes. Successful blockade will be confirmed via a pinprick test prior to transfer to the operating room.

General anesthesia will be induced using intravenous fentanyl (0.5 mcg/kg), propofol (2.5 mg/kg), and rocuronium (0.6 mg/kg). Oral endotracheal intubation will then be performed. Anesthesia will be maintained with sevoflurane (1 MAC) and a continuous remifentanil infusion at a rate of 0.05-0.2 mcg/kg/min. NIBP, HR, and peripheral oxygen saturation will be monitored at 0, 5, 10, and 15 minutes, and every 15 minutes thereafter.

The remifentanil infusion rate will be adjusted based on intraoperative changes in mean arterial pressure (MAP) relative to the preoperative baseline:

* For MAP changes of 10-20%, the dose will be adjusted by ±25%.
* For changes of 20-30%, by ±50%.
* For changes exceeding 30%, by ±50-100%. The goal is to maintain MAP above 60 mmHg and within ±30% of the baseline value.

Thirty minutes prior to extubation, multimodal analgesia will be initiated with 50 mg of intravenous dexketoprofen and 1 g of intravenous paracetamol. During emergence, neuromuscular blockade will be reversed using intravenous neostigmine (0.02 mg/kg) and atropine (0.5 mg). Remifentanil and sevoflurane will be discontinued after surgical dressing, and extubation time will be recorded as the interval between anesthetic discontinuation and endotracheal tube removal.

Intraoperative bleeding will be assessed using the Boezaart Bleeding Score during airway suctioning before extubation (0 = no bleeding, 1 = mild bleeding not requiring suctioning, 2 = mild bleeding requiring occasional suctioning, 3 = mild bleeding requiring frequent suctioning, 4 = moderate bleeding, 5 = severe bleeding).

Total intraoperative remifentanil and sevoflurane consumption, duration of surgery, and total anesthesia time will be recorded. After surgery, patients will be transferred to the post-anesthesia care unit (PACU).

Postoperative pain will be assessed at hour 0 and subsequently at 1, 2, 4, 6, 12, and 24 hours using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain). In accordance with the standard protocol of the otorhinolaryngology department, all patients will receive 50 mg of intravenous dexketoprofen twice daily during the postoperative period. For those requiring additional analgesia (NRS > 4), 1 g of intravenous paracetamol will be administered as rescue medication.

The Quality of Recovery-15 (QoR-15) questionnaire will be re-administered at 24 hours postoperatively and again at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Those with an ASA (American Society of Anesthesiologists) score of I-II
* Those with a body mass index (BMI) between 18 and 30
* Those scheduled for elective surgery
* Those who are fully cooperative Patients who meet the criteria for septorhinoplasty surgery

Exclusion Criteria:

* Conditions that constitute a relative contraindication to regional anesthesia (e.g., coagulation disorders, thrombocytopenia, severe valvular heart disease, local infection at the injection site, allergy to local anesthetic agents)
* International Normalized Ratio (INR) > 1.5
* Facial paralysis or a history of facial paralysis
* History of central nervous system vascular disease
* Presence of neuropathy
* History of surgery in the region where the block will be performed
* American Society of Anesthesiologists (ASA) physical status classification of III or higher
* Patients who do not want to participate in the study
* Patients with chronic pain or chronic opioid use
* Patients with alcohol, substance or drug addiction
* Patients with limited cooperation such as dementia, psychiatric disorders
* Pregnant and breastfeeding patients will be excluded from the study.
* Patients who cannot communicate in their native language will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-11-08 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | İntraoperative-From induction of anesthesia to extubation (anesthesia duration)
  Intraoperative remifentanil infusion will be initiated at 0.05 µg·kg-¹·min-¹. In accordance with the protocol, the rate will be titrated upward or downward based on arterial blood pressure, and the total intraoperative remifentanil dose will be recorded. The average remifentanil dose will be calculated by dividing the total dose by the total anesthesia time and the patient's body weight, and reported as µg·kg-¹·min-¹ and µg·kg-¹·h-¹

SECONDARY OUTCOMES:
Intraoperative sevoflurane consumption | İntraoperative-İntraoperative-From induction of anesthesia to extubation (anesthesia duration)
  At extubation, the anesthesia machine's agent-consumption display will be checked and the total sevoflurane usage recorded. The amount of sevoflurane used for the patient will be documented in milliliters (mL)
Extubation time | From the discontinuation of remifentanil and sevoflurane anesthesia until the time of tracheal extubation, assessed up to 30 minutes post-anesthesia discontinuation
  Following completion of the surgical procedure, administration of remifentanil and sevoflurane anesthesia will be discontinued. The time measurement will start at the moment of discontinuation. The patient will be observed until the return of spontaneous breathing, and the time interval between anesthesia discontinuation and tracheal extubation will be recorded in seconds (s).
Postoperative pain | Postoperative day 1 (0-24 hours)
  Postoperative pain will be assessed at hour 0 and subsequently at 1, 2, 4, 6, 12, and 24 hours using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain).
Anesthesiologist, surgeon and patient satisfaction will be evaluated | Satisfaction ratings for the surgeon and anesthesiologist will be obtained immediately after surgery; the patient will be assessed at 24 hours postoperatively.
  Immediately after surgery, surgeon and anesthesiologist satisfaction will be assessed. At 24 hours postoperatively, the patient will be asked to rate overall perioperative satisfaction. Surgeon, anesthesiologist, and patient satisfaction will be scored on a 5-point Likert scale: 1 = far below expectations; 2 = below expectations; 3 = met expectations; 4 = above expectations; 5 = far above expectations. For all items, the scale will be anchored such that 5 indicates the best score and 1 the worst.
Postoperative bleeding index (Boezaart Bleeding Score) | İntraoperative ( during extubation)
  Boezaart Bleeding Score during airway suctioning before extubation (0 = no bleeding, 1 = mild bleeding not requiring suctioning, 2 = mild bleeding requiring occasional suctioning, 3 = mild bleeding requiring frequent suctioning, 4 = moderate bleeding, 5 = severe bleeding)
The Quality of Recovery-15 (QoR-15) questionnaire | To be examined in the preoperative phase, at the 24th hour postoperatively and at the 1st month postoperatively
  Administration and assessment time points This is a patient-reported outcome measure (PROM). In this study, it will be administered at three time points: (1) preoperative baseline; (2) 24 hours postoperatively; and (3) 1 month postoperatively. Instrument structure and scoring: The instrument comprises 15 items, each rated on a 0-10 numeric scale. Section A (10 items): 0 = never (poor), 10 = always (excellent). Higher scores indicate better well-being. Section B (5 symptom items): 0 = constantly (poor), 10 = never (excellent). The absence of symptoms is reflected by higher scores; therefore, no reverse-coding is required.Total score and interpretation. The total QoR-15 score is obtained by summing all 15 items and ranges from 0 to 150. Lowest possible total score (worst): 0,Highest possible total score (best): 150.

CONTACTS AND LOCATIONS:
Overall Officials: Emine ARIK, Associate Professor, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)